CLINICAL TRIAL: NCT06979297
Title: Promoting Physical Activity and Healthy Eating in Latinas Via Interactive Web-Based Technology
Brief Title: Promoting Physical Activity and Healthy Eating in Latinas
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2022003270; 5K01HL159044 (NIH)
Record Dates: First submitted 2025-05-16; First posted 2025-05-18 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Physical Inactivty; Physical Activity; Diet Quality
Keywords: healthy eating; dietary intervention; lifestyle intervention; physical activity; physical inactivity
MeSH Terms: conditions — Motor Activity; Sedentary Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Web-based physical activity and diet intervention (Experimental)
  Interventions: Behavioral: Web-based physical activity and diet intervention
- Wait-list control arm (Other)
  Interventions: Other: Wait-list control arm

INTERVENTIONS:
Behavioral: Web-based physical activity and diet intervention — Participants receive access to a theory-driven, web-based intervention for 12 weeks that provides interactive information on diet and physical activity, including goal setting, diet and activity tracking, tailored information on healthy eating and increasing exercise, and videos on topics of healthy eating and physical activity.
  Arms: Web-based physical activity and diet intervention
Other: Wait-list control arm — Participants in the wait-list control will complete all the same measures as the intervention group for the first 12 weeks, then will receive access to the Internet-based intervention for another 12 weeks.
  Arms: Wait-list control arm

SUMMARY:
The goal of this clinical trial is to learn if an Internet-based behavioral intervention can increase physical activity and improve diet quality among Latina adults. The main question aims to answer is whether participants in the Internet-based behavioral intervention group increase their physical activity levels, increase their consumption of fruits and vegetables, and decrease their consumption of sugar-sweetened beverages over 12 weeks. Researchers will compare the Internet-based physical activity and healthy eating intervention to a wait-list control group (participants who do not receive any intervention until after completing the study) to see if the Internet-based behavioral intervention works to improve physical activity and diet quality. Participants who receive the Internet-based behavioral intervention receive access to the online intervention for 12 weeks, and complete assessments at baseline and week-12. Participants in the wait-list control complete the same assessments at baseline and week 12, then receive access to the online intervention for 12 weeks.

DETAILED DESCRIPTION:
Participants (N=70) will be Latinas aged 18 years and over who report insufficient physical activity levels, insufficient consumption of fruits and vegetables, and regular consumption of sugar-sweetened beverages (according to the National Guidelines for Physical Activity and National Dietary Guidelines for Americans). Participants who meet eligibility criteria will attend an online orientation session where they will receive thorough information about the study, including any risks/benefits, study requirements and expectations, and will have the opportunity to ask questions about the study. Latinas who are interested in participating will complete the informed consent process and will be mailed an accelerometer with detailed instruction to wear during the next seven days (until their baseline visit). At their online baseline visit, participants will complete physical activity and dietary assessments and will be randomized to one of two study conditions: 1) the PA and Diet Intervention, or 2) the wait-list control. Participants randomized to the PA and Diet Intervention arm will be given access to an interactive Internet-based intervention for 12 weeks, will establish their goals for increasing fruits and vegetables, decreasing sugar-sweetened beverages, and increasing physical activity, and will complete assessments at baseline and 12 weeks. Participants in the wait-list control will complete the same measures as the intervention group for the first 12 weeks, then will receive access to the Internet-based intervention for another 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

Ages 18 years and over; Self-identify as Hispanic or Latino (or of a group defined as Hispanic/Latino by the Census Bureau); Report insufficient PA levels (according to the national PA guidelines); Consume less than 1.5 cups of fruit/day and 2.5 cups of vegetables/day, and/or consume SSB ≥2 times/week; Have regular access to an Internet-connected device through phone, home, work, or their community (e.g., public library, community center, neighbor's house); Are not pregnant or planning to become pregnant during the course of the study.

Exclusion Criteria:

Any orthopedic condition that would limit their mobility; History of heart disease, stroke or any other health condition that would make PA or dietary change unsafe.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-05-28 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Accelerometer-measured min/week moderate to vigorous physical activity (MVPA) | Baseline and 12 weeks
  All participants will wear an Actigraph GT3X+ accelerometer during the week prior to their baseline and week 12 assessments. The Actigraph is a device that measures movement and intensity of activity and has been validated against heart rate telemetry and total energy expenditure.
Consumption of fruit and vegetables | Baseline and 12 weeks
  All participants will complete the NCI Eating at America's Table All Day Fruit and Vegetable Screener at baseline and week 12. The NCI Eating at America's Table Fruit and Vegetable Screener is self-report questionnaire that assesses the frequency of usual fruit and vegetable consumption.
Consumption of sugar-sweetened beverages | Baseline and 12 weeks
  All participants will complete the Beverage Intake Questionnaire (BEV-Q) at baseline and week 12. The BEV-Q is a self-administered, valid and reliable tool measuring the frequency and amount of beverages consumed in 19 categories of drinks, including sugar-sweetened beverages.

CONTACTS AND LOCATIONS:
Locations (1):
- Brown University, Providence, Rhode Island, United States